CLINICAL TRIAL: NCT02207530
Title: A Phase II, Multi-Center, Single-Arm, Global Study of MEDI4736 Monotherapy in Patients With Recurrent or Metastatic Squamous Cell Carcinoma of the Head and Neck (SCCHN)
Brief Title: Phase II Study of MEDI4736 Monotherapy in Treatment of Recurrent or Metastatic Squamous Cell Carcinoma of the Head and Neck
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: PRA Health Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D4193C00001
Record Dates: First submitted 2014-08-01; First posted 2014-08-04 (Estimated); Results first posted 2018-06-18 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Recurrent or Metastatic PD-L1-positive Squamous Cell Carcinoma of the Head and Neck
Keywords: Head and neck cancer; SCCHN
MeSH Terms: conditions — Recurrence; Head and Neck Neoplasms | interventions — durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MEDI4736 (Experimental): MEDI4736 monotherapy
  Interventions: Drug: MEDI4736

INTERVENTIONS:
Drug: MEDI4736 — MEDI4736 monotherapy

SUMMARY:
Primary Objective: To assess the efficacy of MEDI4736 monotherapy in terms of ORR

DETAILED DESCRIPTION:
This is a phase II, multi-center, single-arm, global study of MEDI4736 monotherapy in patients with PD-L1 positive recurrent or metastatic Squamous Cell Carcinoma of the Head and Neck (SCCHN), who have progressed during or after treatment with only 1 systemic palliative regimen for recurrent or metastatic disease that must have contained a platinum agent.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Written informed consent obtained from the patient/legal representative
* Histologically confirmed recurrent or metastatic SCCHN
* Tumor progression or recurrence during or after treatment with only 1 systemic palliative regimen for recurrent or metastatic disease that must have contained a platinum agent.
* Written consent to provide newly acquired tumor tissue (preferred) or archival tissue for the purpose of establishing PD-L1 status.
* Confirmed PD-L1-positive SCCHN by Ventana SP263 assay
* WHO/ECOG performance status of 0 or 1
* At least 1 measurable lesion at baseline
* No prior exposure to immune-mediated therapy
* Adequate organ and marrow function
* Evidence of post-menopausal status or negative urinary or serum pregnancy test.

Exclusion Criteria:

* Histologically confirmed squamous cell carcinoma of any other primary anatomic location in the head and neck
* Received more than 1 systematic palliative regimen for recurrent or metastatic disease
* Any concurrent chemotherapy, Investigational Product, biologic, or hormonal therapy for cancer treatment
* Prior randomization or treatment in a previous MEDI4736 and/or tremelimumab clinical study regardless of treatment arm assignment or receipt of any investigational anticancer therapy within 28 days or 5 half-lives
* Receipt of last dose of an approved (marketed) anticancer therapy (chemotherapy, targeted therapy, biologic therapy, mAbs, etc) within 21 days prior to the first dose of study treatment
* Major surgical procedure within 28 days prior to the first dose of Investigational Product
* Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criterion
* Current or prior use of immunosuppressive medication within 14 days before the first dose of MEDI4736
* History of allogeneic organ transplantation
* Active or prior documented autoimmune or inflammatory disorders;
* Uncontrolled intercurrent illness
* Another primary malignancy
* Patients with history of brain metastases, spinal cord compression, or leptomeningeal carcinomatosis
* History of active primary immunodeficiency
* Known history of previous tuberculosis
* Active infection including hepatitis B, hepatitis C or human immunodeficiency virus (HIV)
* Receipt of live, attenuated vaccine within 30 days prior to the first dose of MEDI4736
* Pregnant or breast-feeding female patients
* Mean QT interval corrected for heart rate (QTc) ≥470 ms calculated from 3 electrocardiograms (ECGs) using Fridericia's Correction
* Any condition that, in the opinion of the Investigator, would interfere with evaluation of the IP or interpretation of patient safety or study results

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2014-10-23 (Actual); Primary Completion 2016-09-26 (Actual); Study Completion 2020-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dan Paul Zandberg, MD, Principal Investigator — International Coordinating Investigator; Magdalena Wrona, Study Director — Medical Scientist AstraZeneca Magdalena.Wrona@astrazeneca.com
Locations (97):
- United States (35):
  - Research Site, Birmingham, Alabama
  - Research Site, Yuma, Arizona
  - Research Site, Duarte, California
  - Research Site, Fullerton, California
  - Research Site, Long Beach, California
  - Research Site, Los Angeles, California
  - Research Site, San Francisco, California
  - Research Site, Whittier, California
  - Research Site, Denver, Colorado
  - Research Site, Jacksonville, Florida
  - Research Site, Augusta, Georgia
  - Research Site, Macon, Georgia
  - Research Site, Evanston, Illinois
  - Research Site, Lexington, Kentucky
  - Research Site, Baltimore, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Southfield, Michigan
  - Research Site, Minneapolis, Minnesota
  - Research Site, Rochester, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, Lebanon, New Hampshire
  - Research Site, Buffalo, New York
  - Research Site, New York, New York
  - Research Site, Stony Brook, New York
  - Research Site, Durham, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Portland, Oregon
  - Research Site, Germantown, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, Fairfax, Virginia
  - Research Site, Morgantown, West Virginia
  - Research Site, Milwaukee, Wisconsin
- Belgium (5):
  - Research Site, Brussels
  - Research Site, Kortrijk
  - Research Site, Leuven
  - Research Site, Montigny-le-Tilleul
  - Research Site, Namur
- Canada (5):
  - Research Site, Calgary, Alberta
  - Research Site, London, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
- Research Site, Zlín, Czechia
- France (17):
  - Research Site, Angers
  - Research Site, Bordeaux
  - Research Site, Brest
  - Research Site, Clermont-Ferrand
  - Research Site, Dijon
  - Research Site, Le Mans
  - Research Site, Lille
  - Research Site, Lorient
  - Research Site, Lyon
  - Research Site, Montpellier
  - Research Site, Nice
  - Research Site, Plerin SUR MER
  - Research Site, Rouen
  - Research Site, Saint-Grégoire
  - Research Site, Strasbourg
  - Research Site, Toulouse
  - Research Site, Villejuif
- Georgia (2):
  - Research Site, Batumi
  - Research Site, Tbilisi
- Germany (5):
  - Research Site, Berlin
  - Research Site, Halle
  - Research Site, Heidelberg
  - Research Site, Leipzig
  - Research Site, München
- Hungary (2):
  - Research Site, Budapest
  - Research Site, Gyula
- Israel (3):
  - Research Site, Haifa
  - Research Site, Petah Tikva
  - Research Site, Tel Litwinsky
- Malaysia (3):
  - Research Site, Kuala Lumpur
  - Research Site, Kuching
  - Research Site, Sabak Bernam
- South Korea (4):
  - Research Site, Daegu
  - Research Site, Goyang-si
  - Research Site, Seoul
  - Research Site, Suwon
- Spain (9):
  - Research Site, Barakaldo
  - Research Site, Barcelona
  - Research Site, L'Hospitalet de Llobregat
  - Research Site, Madrid
  - Research Site, Marbella (Málaga)
  - Research Site, Málaga
  - Research Site, Pamplona
  - Research Site, Valencia
  - Research Site, Zaragoza
- Research Site, Taipei, Taiwan
- United Kingdom (5):
  - Research Site, Birmingham
  - Research Site, Glasgow
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Metropolitan Borough of Wirral

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 110 sites in 14 countries enrolled and screened patients. The study was conducted and managed by PRA, a contract research organization.
Groups:
- MEDI4736 10 mg/kg: MEDI4736 monotherapy: Durvalumab was provided at a dose of 10 mg/kg using an intravenous solution every 2 weeks until 12 months, disease progression, toxicity, or patient decision to stop therapy
Period: Overall Study
Arm/Group | MEDI4736 10 mg/kg
Started | 112
Completed | 21
Not Completed | 91
Not completed — Worsening condition under investigation | 78
Not completed — Patient decision to stop study treatment | 5
Not completed — Adverse Event | 8

BASELINE CHARACTERISTICS:
Population: Full analysis set - included all treated patients who had a baseline tumor assessment and had measurable disease at baseline according to the Investigator site assessment.
Arm/Group | MEDI4736 10 mg/kg
Number analyzed (Participants) | 112
Age, Categorical [Count of Participants; unit: Participants] — Population: Full analysis set - included all treated patients who had a baseline tumor assessment and had measurable disease at baseline according to the Investigator site assessment.
  Participants
    <=18 years | 0
    Between 18 and 65 years | 83
    >=65 years | 29
Age, Continuous [Median (Full Range); unit: Years] — Population: Full analysis set - included all treated patients who had a baseline tumor assessment and had measurable disease at baseline according to the Investigator site assessment.
  Years | 60.0 [24 to 84]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Full analysis set - included all treated patients who had a baseline tumor assessment and had measurable disease at baseline according to the Investigator site assessment.
  Participants
    Female | 32
    Male | 80
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Full analysis set - included all treated patients who had a baseline tumor assessment and had measurable disease at baseline according to the Investigator site assessment.
  Participants
    Hispanic or Latino | 1
    Not Hispanic or Latino | 109
    Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Full analysis set - included all treated patients who had a baseline tumor assessment and had measurable disease at baseline according to the Investigator site assessment.
  Participants
    American Indian or Alaska Native | 0
    Asian | 4
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 5
    White | 100
    More than one race | 0
    Unknown or Not Reported | 3
Smoking/ Nicotine status [Number; unit: Participants] — Population: Full analysis set - included all treated patients who had a baseline tumor assessment and had measurable disease at baseline according to the Investigator site assessment.
  Participants
    >10 Pack years | 49
    <=10 pack years | 53
    Unknown/ Not reported | 10
Nicotine Use [Number; unit: Participants] — Population: Full analysis set - included all treated patients who had a baseline tumor assessment and had measurable disease at baseline according to the Investigator site assessment.
  Participants
    Current | 10
    Former | 59
    Never | 43
HPV status [Number; unit: Participants] — Population: Full analysis set - included all treated patients who had a baseline tumor assessment and had measurable disease at baseline according to the Investigator site assessment.
  Participants
    Positive | 34
    Negative | 65
    Unknown/ Not reported | 3
WHO/ECOG performance status [Number; unit: Participants] — Population: Full analysis set - included all treated patients who had a baseline tumor assessment and had measurable disease at baseline according to the Investigator site assessment.
  Participants
    (0) Normal activity | 34
    (1) Restricted activity | 77
    Missing | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: Objective response rate (per RECIST 1.1 as assessed by blinded independent central review [BICR]) is defined as the number (%) of patients with a confirmed complete response or confirmed partial response and will be based on all treated patients who are PD-L1-positive with measurable disease at baseline per BICR.
  Response Evaluation Criteria in Solid Tumors [RECIST] 1.1. criteria are: Complete response [CR] = disappearance of all target lesions since baseline; and partial response [PR] = at least a 30% decrease in the sum of the diameters of target lesions.
Time Frame: 12 months
Population: Evaluable analysis set - all patients who received at least one dose of study treatment, who had a baseline tumor assessment, and had measurable disease at baseline according to BICR
Measure: Number (95% Confidence Interval); unit: % of participants
Arm/Group | MEDI4736 10 mg/kg
Number analyzed (Participants) | 111
% of participants
  Overall | 16.2 [9.9 to 24.41]
  Smoking/nicotine status >10 pack years: number analyzed (Participants) | 48
  Smoking/nicotine status >10 pack years | 14.6 [6.07 to 27.76]
  Smoking/nicotine status <=10 pack years: number analyzed (Participants) | 53
  Smoking/nicotine status <=10 pack years | 18.9 [9.44 to 31.97]
  Smoking/nicotine status - Missing: number analyzed (Participants) | 10
  Smoking/nicotine status - Missing | 10.0 [NA to NA] — Only 1 patient in this category with a response
  Substance user-Current: number analyzed (Participants) | 9
  Substance user-Current | 11.1 [0.28 to 48.25]
  Substance user-Former: number analyzed (Participants) | 59
  Substance user-Former | 15.3 [7.22 to 26.99]
  Substance user-Never: number analyzed (Participants) | 43
  Substance user-Never | 18.6 [8.39 to 33.40]
  HPV status-Positive: number analyzed (Participants) | 34
  HPV status-Positive | 29.4 [15.10 to 47.48]
  HPV status-Negative: number analyzed (Participants) | 64
  HPV status-Negative | 10.9 [4.51 to 21.25]
  HPV status-Missing: number analyzed (Participants) | 13
  HPV status-Missing | 7.7 [NA to NA] — Only 1 patient in this category with a response

2. Secondary Outcome: Best Objective Response
Description: Best objective response based on BICR assessments according to RECIST v1.1. Response required confirmation after 4 weeks.
  Unconfirmed complete (CR) or partial response (PR) refers to CR or PR achieved but either no confirmation assessment was performed or a confirmation assessment was performed but response was not confirmed.
Time Frame: 12 months
Population: Evaluable analysis set - included all patients who received at least one dose of study treatment who had a baseline tumor assessment and had measurable disease at baseline according to BICR.
Measure: Number; unit: % of participants
Arm/Group | MEDI4736 10 mg/kg
Number analyzed (Participants) | 111
% of participants
  Response-Total | 16.2
  Response-Partial response (PR) | 15.3
  Response-Complete response (CR) | 0.9
  Non-response (NR)-Total | 83.8
  NR-Stable disease (SD)≥8 weeks-Total | 9.0
  NR-SD≥8 weeks-Unconfirmed CR or PR | 2.7
  NR-Stable disease (SD) ≥8 weeks-SD | 6.3
  NR-Progression-Total | 52.3
  NR-Progression-RECIST 1.1 progression | 25.2
  NR-Progression-Death | 27.0
  NR-Not evaluable-Total | 22.5
  NR-Not evaluable-SD<8 weeks | 19.8
  NR-Not evaluable-Incomplete post-baseline tests | 2.7

3. Secondary Outcome: Duration of Response- Participants Remaining in Response
Description: Participants remaining in response - based on BICR assessments according to RECIST v1.1.
  An ongoing response was defined as a patient who had documented objective response and was still alive and progression-free at the time of the data cut-off.
Time Frame: 12 months
Population: as for outcome 2
Measure: Number; unit: % of participants
Arm/Group | MEDI4736 10 mg/kg
Number analyzed (Participants) | 18
% of participants
  Remaining in response-3 months | 100
  Remaining in response-6 months | 76.5
  Remaining in response-9 months | 61.8
  Remaining in response-12 months | 37.1
  Ongoing response | 55.6

4. Secondary Outcome: Duration of Response
Description: Duration of objective response in patients with objective response based on BICR assessments according to RECIST v1.1.
  Duration of response was the time from the first documentation of complete or partial response until the date of progression (which was subsequently confirmed), death, or the last evaluable RECIST assessment for patients that did not progress.
  An ongoing response was defined as a patient who had documented objective response and was still alive and progression-free at the time of the data cut-off.
Time Frame: 12 months
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | MEDI4736 10 mg/kg
Number analyzed (Participants) | 18
Participants
  No. progressed or died within 12 months | 6
  No. progressed or died after 12 months | 2

5. Secondary Outcome: Time to Onset of Response From First Dose
Description: Time to onset of response in patients with objective response based on BICR assessments according to RECIST 1.1
Time Frame: 12 months
Population: as for outcome 2
Measure: Median (Full Range); unit: Months
Arm/Group | MEDI4736 10 mg/kg
Number analyzed (Participants) | 18
Months | 2.00 [1.64 to 9.20]

6. Secondary Outcome: Disease Control at 6 Months
Description: Disease control (DCR) at 6 months based on BICR assessments according to RECIST v1.1.
  DCR at 6 months was evaluated using 2 different approaches to the length of stable disease (SD):
  * Method 1: Patients who had a best objective response of complete response (CR) or partial response (PR) within 24 weeks or had demonstrated SD for a minimum interval of 24 weeks following the start of study treatment.
  * Method 2: Patients who had a best objective response of CR or PR within 24 weeks or had demonstrated SD for a minimum interval of 16 weeks following the start of study treatment.
Time Frame: 6 months
Population: as for outcome 2
Measure: Number; unit: % of participants
Arm/Group | MEDI4736 10 mg/kg
Number analyzed (Participants) | 111
% of participants
  METHOD 1: Disease control at 6 months | 23.4
  METHOD 1: No disease control at 6 months | 76.6
  METHOD 1: No disease control:Not evaluable/missing | 27.0
  METHOD 2: Disease control at 6 months | 33.3
  METHOD 2: No disease control at 6 months | 66.7
  METHOD 2: No disease control:Not evaluable/missing | 27.0

7. Secondary Outcome: Progression-free Survival
Description: Progression status based on BICR assessments according to RECIST v1.1 at time of PFS analysis.
  Progression was defined as the time from the date of first dose until the date of objective disease progression or death (by any cause in the absence of progression) regardless of whether the patient withdrew from therapy or received another anti-cancer therapy prior to progression.
Time Frame: 12 months
Population: as for baseline characteristics
Measure: Number; unit: % of participants
Arm/Group | MEDI4736 10 mg/kg
Number analyzed (Participants) | 112
% of participants
  No progression | 17.0
  No progression + under follow-up | 12.5
  Progression-Total | 83.0
  RECIST 1.1 progression | 50.0
  Death in absence of RECIST 1.1 progression | 33.0

8. Secondary Outcome: Overall Survival (OS)
Description: Survival status at time of overall survival analysis. 'Still in survival follow-up' includes patients known to be alive at data cut-off. 'Terminated prior to death' includes patients with unknown survival status, or who were lost to follow-up.
Time Frame: 12 months
Population: as for baseline characteristics
Measure: Number; unit: % of participants
Arm/Group | MEDI4736 10 mg/kg
Number analyzed (Participants) | 112
% of participants
  Still in survival follow-up | 24.1
  Terminated prior to death | 6.3
  Voluntary discontinuation by subject | 6.3
  Death | 69.6

9. Secondary Outcome: Quality of Life
Description: Improvement in quality of life was assessed using European Organisation for Research and Treatment of Cancer (EORTC) questionnaires:
  * The impact of treatment on Health-Related Quality of Life, functioning, and symptoms was evaluated using the EORTC QLQ-C30 v3.
  * Head and neck cancer-specific symptoms were evaluated using the EORTC QLQ-H&N35.
  Function or global health status/quality of life improvement was defined as patients with 2 consecutive assessments at least 14 days apart that showed a clinically meaningful improvement (an increase from baseline score ≥10). Symptom improvement was defined as 2 consecutive assessments at least 14 days apart that showed a clinically meaningful improvement (a decrease from baseline score ≥10).
  Scale improvement was defined as patients with 2 consecutive assessments at least 14 days apart that showed a clinically meaningful improvement (a decrease from baseline score ≥10).
Time Frame: 12 months
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: % of participants
Arm/Group | MEDI4736 10 mg/kg
Number analyzed (Participants) | 112
% of participants
  EORTC QLQ-C30 Function-Physical: number analyzed (Participants) | 70
  EORTC QLQ-C30 Function-Physical | 17.1 [10.1 to 27.6]
  EORTC QLQ-C30 Function-Role: number analyzed (Participants) | 70
  EORTC QLQ-C30 Function-Role | 22.9 [14.6 to 34.0]
  EORTC QLQ-C30 Function-Cognitive: number analyzed (Participants) | 62
  EORTC QLQ-C30 Function-Cognitive | 21.0 [12.7 to 32.6]
  EORTC QLQ-C30 Function-Emotional: number analyzed (Participants) | 69
  EORTC QLQ-C30 Function-Emotional | 15.9 [9.1 to 26.3]
  EORTC QLQ-C30 Function-Social: number analyzed (Participants) | 75
  EORTC QLQ-C30 Function-Social | 34.7 [24.9 to 45.9]
  EORTC QLQ-C30 Symptom-Fatigue: number analyzed (Participants) | 89
  EORTC QLQ-C30 Symptom-Fatigue | 21.3 [14.1 to 31.0]
  EORTC QLQ-C30 Symptom-Pain: number analyzed (Participants) | 82
  EORTC QLQ-C30 Symptom-Pain | 26.8 [18.4 to 37.3]
  EORTC QLQ-C30 Symptom-Nausea/vomiting: number analyzed (Participants) | 31
  EORTC QLQ-C30 Symptom-Nausea/vomiting | 32.3 [18.6 to 49.9]
  EORTC QLQ-C30 Global health status/QoL: number analyzed (Participants) | 96
  EORTC QLQ-C30 Global health status/QoL | 13.5 [8.1 to 21.8]
  EORTC QLQ-H&N35 Scale-Pain in the mouth: number analyzed (Participants) | 69
  EORTC QLQ-H&N35 Scale-Pain in the mouth | 24.6 [16.0 to 36.0]
  EORTC QLQ-H&N35 Scale-Swallowing: number analyzed (Participants) | 62
  EORTC QLQ-H&N35 Scale-Swallowing | 19.4 [11.4 to 30.9]
  EORTC QLQ-H&N35 Scale-Senses: number analyzed (Participants) | 67
  EORTC QLQ-H&N35 Scale-Senses | 34.3 [24.1 to 46.3]
  EORTC QLQ-H&N35 Scale-Speech: number analyzed (Participants) | 81
  EORTC QLQ-H&N35 Scale-Speech | 28.4 [19.7 to 39.0]
  EORTC QLQ-H&N35 Scale-Social eating: number analyzed (Participants) | 67
  EORTC QLQ-H&N35 Scale-Social eating | 22.4 [14.1 to 33.7]
  EORTC QLQ-H&N35 Scale-Social contact: number analyzed (Participants) | 58
  EORTC QLQ-H&N35 Scale-Social contact | 17.2 [9.6 to 28.9]
  EORTC QLQ-H&N35 Scale-Sexuality: number analyzed (Participants) | 74
  EORTC QLQ-H&N35 Scale-Sexuality | 25.7 [17.1 to 36.7]

ADVERSE EVENTS:
Time Frame: From the time the informed consent was signed through 90 days after the last dose of the last study treatment or until another therapy was initiated.
Description: AEs were reported spontaneously or in response to open questions, revealed by observation, or were changes from baseline/deterioration in tests and vital signs that met SAE criteria or led to IP discontinuation.
  AEs/SAEs were followed up for resolution after discontinuation or study completion and for as long as medically indicated.
Arm/Group | MEDI4736 10 mg/kg
All-Cause Mortality (participants affected / at risk) | 78/112
Serious Adverse Events (participants affected / at risk) | 43/112
Other Adverse Events (participants affected / at risk) | 93/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MEDI4736 10 mg/kg (N=112)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Cardiac arrest (Cardiac disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 1 (1)
Hypercalcaemia of malignancy (Endocrine disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Mouth haemorrhage (Gastrointestinal disorders) | 1 (1)
Oesophageal haemorrhage (Gastrointestinal disorders) | 1 (1)
Pneumatosis intestinalis (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Fatigue (General disorders) | 3 (4)
Localised oedema (General disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 1 (1)
Hepatotoxicity (Hepatobiliary disorders) | 1 (1)
Abscess neck (Infections and infestations) | 1 (1)
Device related infection (Infections and infestations) | 1 (1)
Gangrene (Infections and infestations) | 1 (3)
Gastrointestinal infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 4 (5)
Pulmonary sepsis (Infections and infestations) | 1 (1)
Septic shock (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Gastrostomy failure (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Wound haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2)
Cerebral infarction (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1)
Nerve compression (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Vascular encephalopathy (Nervous system disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Nephritis (Renal and urinary disorders) | 1 (1)
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung cyst (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Stridor (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (2)
Superior vena cava syndrome (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MEDI4736 10 mg/kg (N=112)
Anaemia (Blood and lymphatic system disorders) | 18 (19)
Hypothyroidism (Endocrine disorders) | 15 (15)
Constipation (Gastrointestinal disorders) | 22 (27)
Diarrhoea (Gastrointestinal disorders) | 16 (28)
Dysphagia (Gastrointestinal disorders) | 11 (11)
Nausea (Gastrointestinal disorders) | 22 (28)
Vomiting (Gastrointestinal disorders) | 13 (19)
Asthenia (General disorders) | 17 (18)
Fatigue (General disorders) | 26 (27)
Localised oedema (General disorders) | 6 (6)
Mucosal inflammation (General disorders) | 6 (6)
Pyrexia (General disorders) | 10 (15)
Nasopharyngitis (Infections and infestations) | 7 (10)
Urinary tract infection (Infections and infestations) | 10 (10)
Gamma-glutamyltransferase increased (Investigations) | 7 (7)
Weight decreased (Investigations) | 13 (13)
Decreased appetite (Metabolism and nutrition disorders) | 18 (21)
Hypercalcaemia (Metabolism and nutrition disorders) | 10 (10)
Hypokalaemia (Metabolism and nutrition disorders) | 7 (9)
Hypomagnesaemia (Metabolism and nutrition disorders) | 10 (15)
Hyponatraemia (Metabolism and nutrition disorders) | 8 (14)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (15)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (7)
Neck pain (Musculoskeletal and connective tissue disorders) | 6 (6)
Dizziness (Nervous system disorders) | 11 (13)
Headache (Nervous system disorders) | 10 (14)
Insomnia (Psychiatric disorders) | 10 (12)
Cough (Respiratory, thoracic and mediastinal disorders) | 12 (13)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 15 (18)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Dry skin (Skin and subcutaneous tissue disorders) | 8 (8)
Pruritus (Skin and subcutaneous tissue disorders) | 12 (14)
Rash (Skin and subcutaneous tissue disorders) | 7 (7)
Hypotension (Vascular disorders) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review publications prior to public release for a period up to 120 days to confirm accuracy, prevent disclosure of confidential information, and ensure that information is handled appropriately.